CLINICAL TRIAL: NCT00398294
Title: An Open-Label, Single-Arm, Prospective Study to Evaluate the Lipid-Lowering Efficacy and Safety of Simvastatin 40 Mg Tablet in Patients With Hypercholesterolemia
Brief Title: To Evaluate the Lipid-Lowering Efficacy and Safety of Simvastatin 40 Mg Tablet In Patients With Hypercholesterolemia (0733-264)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0733-264; 2006_044
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Simvastatin; Duration of Therapy

INTERVENTIONS:
Drug: MK0733, simvastatin / Duration of Treatment: 12 Weeks

SUMMARY:
To collect lipid-lowering response data with the use of simvastatin 40 mg tablet in patients with hypercholesterolemia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, >18 years of age
* Patients with hypercholesterolemia who meet the following lipid criteria:

  1. primary cholesterolemia: total cholesterol>=240 mg/dl or ldl-c >= 160 mg/dl
  2. secondary cholesterolemia (patients with cad, dm): ldl-c>=130 mg/dl
* The patient is willing to follow an NCEP therapeutic lifestyle changes (tlc) or similar cholesterol-lowering diet throughout the duration of the study

Exclusion Criteria:

* Congestive heart failure (NYHA class III or IV), uncontrolled cardiac arrhythmias, unstable angina pectoris
* Myocardial infarction, coronary artery bypass surgery, or angioplasty within 3 months of visit 1
* Uncontrolled hypertension with systolic blood pressure > 160 mmhg or diastolic > 100 mmhg at visit 1.
* Unstable diabetes (hba1c >9%) or newly diagnosed (within 3 months)or change in anti-diabetes medications within 3 months of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05-01 (Actual); Primary Completion 2006-04-04 (Actual); Study Completion 2006-04-04 (Actual)

PRIMARY OUTCOMES:
Total cholesterol, ldl-c, hdl-c, and triglycerides after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Merck Sharp & Dohme (I.A.) Corp., Taipei, Taiwan